CLINICAL TRIAL: NCT01152853
Title: A Phase II Open Label Trial of PF-00299804 Monotherapy in Patients With HER-2 Positive Advance Gastric Cancer After Failure of At Least One Prior Chemotherapy Regimen
Brief Title: PF-00299804 Monotherapy in Patients With HER-2 Positive Advance Gastric Cancer
Acronym: PF299804-AGC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-1004-031-315
Record Dates: First submitted 2010-06-20; First posted 2010-06-29 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-05

CONDITIONS: Advanced Gastric Cancer; HER2
Keywords: advanced gastric cancer; HER2; PF00299804
MeSH Terms: interventions — dacomitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- single arm (Experimental): PF00299804 treatment arm
  Interventions: Drug: PF00299804

INTERVENTIONS:
Drug: PF00299804 — PF-00299804 will be given orally once daily at 45 mg daily. Patients will take study drug continuously, with cycles of 28 days.
  Other Names: PF-00299804

SUMMARY:
In case of gastric cancer, the incidence of HER-2 positivity (2+, 3+ on IHC and/or FISH (+)) is reported as similar as that of breast cancer, that is 22% of all cases. A recent ToGA Trial, phase III trial comparing trastuzumab combined with chemotherapy (fluoropyrimidine+cisplatin) versus chemotherapy alone in chemotherapy-naïve HER-2 (+) gastric cancer shows the significant benefit of using trastuzumab in terms of overall survival and progression-free survival. It provides the clinical evidence of HER-2 as a reasonable and potential therapeutic target in gastric cancer.

Nowadays, lapatinib, HER-1 and HER-2 dual inhibitor, is also testing under the clinical trial in gastric cancer.

In preclinical study, PF-00299804 is highly active in HER-2 amplified gastric cancer cell lines.(SNU preclinical data) So, we plan this phase II trial of PF-00299804 monotherapy in patients with HER-2 positive advance gastric cancer after failure of at least one chemotherapy regimen.

DETAILED DESCRIPTION:
The role of HER-2 during carcinogenesis and its prognostic role in breast cancer has been already well established. Furthermore the value of HER-2 as a reasonable therapeutic target in breast cancer has translated into the good clinical therapeutic result using HER-2 targeting agent, such as trastuzumab and lapatinib.

In case of gastric cancer, the incidence of HER-2 positivity (2+, 3+ on IHC and/or FISH (+)) is reported as similar as that of breast cancer, that is 22% of all cases. A recent ToGA Trial, phase III trial comparing trastuzumab combined with chemotherapy (fluoropyrimidine+cisplatin) versus chemotherapy alone in chemotherapy-naïve HER-2 (+) gastric cancer shows the significant benefit of using trastuzumab in terms of overall survival and progression-free survival. It provides the clinical evidence of HER-2 as a reasonable and potential therapeutic target in gastric cancer.

Nowadays, lapatinib, HER-1 and HER-2 dual inhibitor, is also testing under the clinical trial in gastric cancer.

PF-00299804 is an orally available, potent, and highly selective irreversible small molecule inhibitor of the Human Epidermal Growth Factor Receptor (HER) family of tyrosine kinases:HER-1 (EGFR), HER-2 and HER-4 (HER-3 does not possess kinase activity). PF-00299804 inhibits the tyrosine kinase activity of the HER family through binding at the ATP binding site, which results in covalent modification of a cystine in the ATP binding pocket. The unique irreversible and highly selective properties of PF-00299804 for the HER kinase family results in sustained suppression of receptor tyrosine kinase activity. The long-lasting inhibition of receptor phosphorylation reduces concern over potentially short plasma half-lives. Furthermore, the low nanomolar potency and irreversible binding of the intended targets reduce the need for high peak plasma levels, which in turn could minimize target-nonspecific toxicities.

In preclinical study, PF-00299804 is highly active in HER-2 amplified gastric cancer cell lines.(SNU preclinical data)

Overall, the standard of care for advanced gastric cancer has been of modest benefit with plateau in response rates using various combination chemotherapies. Therefore, development of treatment options for these advanced gastric cancer patients, especially HER-2 (+) gastric cancer patients, remains a target of active research.

So, the investigators plan this phase II trial of PF-00299804 monotherapy in patients with HER-2 positive advance gastric cancer after failure of at least one chemotherapy regimen.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* A patient who is able to walk and should have ECOG performance status of 0-2.
* Histologically confirmed adenocarcinoma of the stomach or gastro-oesophageal junction with inoperable locally advanced or recurrent and/or metastatic disease, not amenable to curative therapy.
* HER2 positive tumour (primary tumour or metastasis defined as 1) 3+ on IHC and/or 2) FISH (+)
* Failure to at least one chemotherapy regimen

  * trastuzumab or lapatinib-pretreated patient is eligible
* Measurable or non-measurable-evaluable disease according to the Response Evaluation Criteria in Solid Tumors (RECIST)
* Adequate bone marrow function, including:
* Adequate renal function, including:
* Adequate liver function, including:
* Adequate Cardiac Function, including:

  1. 12-Lead electrocardiogram (ECG) with normal tracing or non-clinically significant changes that do not require medical intervention;
  2. QTc interval 470 msec and without history of Torsades de Pointes or other symptomatic QTc abnormality;
  3. LVEF (by MUGA or echocardiogram) of ≥50%.
* Brain metastasis allowed if any necessary treatment has been completed and the patient is radiologically and neurologically stable off corticosteroids at least 2 weeks prior to enrollment
* A patient with the willingness to comply with the study protocol during the study period and capable of complying with it.
* A patient who signed the informed consent prior to the participation of the study and who understands that he/she has a right to withdrawal from participation in the study at any time without any disadvantages.

Exclusion Criteria:

* Patients with known active brain metastases or any leptomeningeal metastases;

  a. Patients with previously diagnosed brain metastases for which treatment (radiation or surgery) is recommended in judgment of investigator are eligible if they have completed their CNS treatment and have recovered from the acute effects of radiation therapy or surgery prior to the start of study medication, have discontinued corticosteroid treatment for these metastases for at least 2 weeks and are neurologically stable.
* Radiotherapy (other than palliative radiotherapy to lesions that will not be followed for tumor assessment on this study, ie, non-target lesions), biological or investigational agents within 2 weeks of baseline disease assessments
* Any surgery (not including minor procedures) within 4 weeks of baseline disease assessments; or not fully recovered from any side effects of previous procedures;
* Any clinically significant gastrointestinal abnormalities, which may impair intake, transit or absorption of the study drug, such as the inability to take oral medication in tablet form;
* Current enrollment in another therapeutic clinical trial;
* Any psychiatric or cognitive disorder that would limit the understanding or rendering of informed consent and/or compromise compliance with the requirements of this protocol
* Patients with known interstitial lung disease;
* Uncontrolled or significant cardiovascular disease
* Prior malignancy: Patients will not be eligible if they have evidence of other malignancy (other than non-melanoma skin cancer or in situ cervical cancer, or localized and presumed cured prostate cancer with PSA < ULN) within the last 5 years.
* Organ allogenic transplantation requiring immunosuppressive therapy.
* A patient who developed uncontrolled serious infection or other uncontrolled serious concomitant diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-07; Primary Completion 2011-07 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
progression-free survival at 4-months (PFS4mo) | 10 months
  PFS is defined as the interval from the date of enrollment to the date of disease progression or death due to any cause, whichever occurs first. PFS4m is defined as the proportion of patients alive and progression-free at 4 months relative to all enrolled patients.

SECONDARY OUTCOMES:
Overall Response Rate | 6 months
  Overall Response Rate (BOR) per RECIST Confirmed responses are defined as those that persist on a follow-up imaging assessment 4 weeks after the initial objective documentation of response.
Overall Survival (OS) | 2 years
  Overall Survival (OS), defined as the time from enrollment to the date of death due to any cause.
toxicity | 12 months
  Overall Safety Profile, as characterized by type, frequency, severity as graded by NCI Common Toxicity Criteria for Adverse Events version 3.0 (NCI CTCAEv3.0), timing and relationship to treatment, and laboratory abnormalities observed.

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Jue Bang, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Oh DY, Lee KW, Cho JY, Kang WK, Im SA, Kim JW, Bang YJ. Phase II trial of dacomitinib in patients with HER2-positive gastric cancer. Gastric Cancer. 2016 Oct;19(4):1095-1103. doi: 10.1007/s10120-015-0567-z. Epub 2015 Nov 18. PMID 26581547